CLINICAL TRIAL: NCT01564459
Title: A Phase IIa, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial to Evaluate the Safety and Efficacy of MK-6096 in Patients With Painful Diabetic Neuropathy
Brief Title: Study to Evaluate MK-6096 in the Treatment of Painful Diabetic Neuropathy (PDN) in Adults (MK-6096-021)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6096-021
Record Dates: First submitted 2012-02-28; First posted 2012-03-27 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — MK-6096

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- MK-6096 10 mg→MK-6096 10 mg (Experimental): Participants receive MK-6096 10 mg during run-in once daily for 1 week and receive MK-6096 10 mg once daily for 2 weeks during double-blind treatment period.
  Interventions: Drug: MK-6096
- MK-6096→Placebo (Placebo Comparator): Participants receive MK-6096 10 mg during run-in once daily for 1 week and receive placebo once daily for 2 weeks during double-blind treatment period.
  Interventions: Drug: MK-6096; Drug: Placebo

INTERVENTIONS:
Drug: MK-6096 — MK-6096 10 mg compressed tablets, taken once daily at bedtime for 14 days.
Drug: Placebo — Matching compressed tablets, taken once daily at bedtime for 14 days.
  Arms: MK-6096→Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of MK-6096 in the treatment of painful diabetic neuropathy (PDN) in adults.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of painful diabetic neuropathy (PDN) for at least 6 months.
* Is able to understand & use an electronic diary to complete daily questionnaires.
* If female of reproductive potential, agrees to use acceptable contraception from Screening through to at least 2 weeks after last dose of study drug.
* Is on a stable dose of antihyperglycemic treatment for at least 1 month, with hemoglobin A1C level of no more than 11%.
* If taking an allowable around-the-clock medication for chronic pain, has been on a stable dose for at least 1 month & agrees to stay on same dose during the study.
* Agrees to not start therapy with opioids, pregabalin, gabapentin, duloxetine or any other medications used to treat neuropathic pain during the study.
* Has a regular bedtime of before 1 AM (01:00).
* Agrees to limit alcohol consumption to no more than 3 drinks a day, with no drinks within 3 hours before bedtime. One drink is defined as: 1) 12 ounces of beer; 2) 4 ounces of wine; or 3) 1 ounce of liquor (80 proof or 40% alcohol).
* Agrees to limit caffeine consumption to no more than 5 standard 6-oz. cups of caffeinated beverages or no more than 600 mg caffeine a day, with no caffeinated beverages after 4 PM (16:00).
* Agrees to maintain a relatively consistent level of activity throughout the study.

Exclusion Criteria:

* Is pregnant or breastfeeding, or expects to become pregnant during the study.
* Expects to donate eggs or sperm during the study or within 90 days after last dose of study drug.
* Has had ineffective treatment with more than 3 neuropathic pain drugs.
* Anticipates need for surgery during the study.
* Has another existing type of pain that is as severe as or greater than the pain under study OR is not able to distinguish the pain under study from another existing pain condition.
* Has post herpetic neuralgia (PHN); small fiber predominant neuropathy (SFN); idiopathic sensory neuropathy (ISN); complex regional pain syndrome; sensory neuropathies; or pain caused by radiation/chemotherapy/amputation/human immunodeficiency virus (HIV) infection.
* Has received a nerve block for pain within past 6 weeks.
* Has a history of pernicious anemia, untreated hypothyroidism, or amputations other than toes.
* Has a history of narcolepsy, cataplexy, circadian rhythm disorder, parasomnia, sleep-related breathing disorder, restless legs syndrome, periodic limb movement disorder, excessive daytime sleepiness, or difficulty sleeping due to a medical condition (i.e. asthma, Gastroesophageal Reflux Disease (GERD)) other than PDN.
* Has any history of a neurological disorder, including: seizure disorder, stroke, transient ischemic attack, multiple sclerosis, cognitive impairment, or significant head trauma with sustained loss of consciousness.
* Has a current evidence or history within past 6 months of unstable cardiovascular disorder, including: acute coronary syndrome; unstable angina; congestive heart failure; cardiogenic syncope; cardiomyopathy; or symptomatic arrhythmia.
* Has a Body Mass Index (BMI) of more than 40 kg/m^2.
* Has any of the following: 1) evidence of ongoing depression or suicidality; 2) a lifetime history of bipolar disorder, a psychotic disorder, or posttraumatic stress disorder; 3) a psychiatric condition requiring treatment with a prohibited medication; or 3) other current psychiatric condition that might interfere with ability to participate in the study.
* Is at imminent risk of self-harm or harm to others.
* Has a history of substance abuse or dependence. Substances include alcohol, marijuana, hypnotics, other prescription drugs, & drugs of abuse, but exclude nicotine.
* Has a history of malignant cancer within past 5 years, except for adequately treated basal cell or squamous cell skin cancer or cervical cancer.
* Has a history of hypersensitivity or reaction to more than 2 chemical classes of drugs, including prescription & over-the-counter medications.
* Is currently participating or has participated in an investigational study of a compound or device within past 30 days OR is not willing to refrain from participating in another study during this study.
* Has a history of travel across 3 or more time zones or shift work (permanent night shift or rotating day/night shift work) within past 2 weeks, OR anticipates need to travel across 3 or more time zones during the study.
* Has donated blood products or had more than 300 mL of blood drawn within past 8 weeks; has received blood products within past 30 days; OR intends to donate or receive blood products during the study.
* Has previously participated in a study of MK-6096.
* Is an employee and/or a family member of one of the investigators, study staff, or Merck.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2013-04-18 (Actual); Study Completion 2013-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Joseph Herring W, Ge JY, Jackson S, Assaid C, Connor KM, Michelson D. Orexin Receptor Antagonism in Painful Diabetic Neuropathy: A Phase 2 Trial With Filorexant. Clin J Pain. 2018 Jan;34(1):37-43. doi: 10.1097/AJP.0000000000000503. PMID 28448426

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-6096 10 mg→No Treatment: Participants who received MK-6096 10 mg during run-in and did not continue to double-blind treatment period.
- MK-6096 10 mg→MK-6096 10 mg: Participants that received MK-6096 10 mg during run-in and were randomly assigned to receive MK-6096 10 mg during double-blind treatment period.
- MK-6096 10 mg→Placebo: Participants that received MK-6096 10 mg during run-in and were randomly assigned to receive placebo during double-blind treatment period.
Period: Run-In
Arm/Group | MK-6096 10 mg→No Treatment | MK-6096 10 mg→MK-6096 10 mg | MK-6096 10 mg→Placebo
Started | 12 | 87 (1 participant randomized to placebo arm received MK-6096 10 mg) | 83 (1 participant randomized to placebo arm received MK-6096 10 mg)
Completed | 0 | 87 | 83
Not Completed | 12 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-compliance with study drug | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Double-blind Treatment
Arm/Group | MK-6096 10 mg→No Treatment | MK-6096 10 mg→MK-6096 10 mg | MK-6096 10 mg→Placebo
Started | 0 | 87 (1 participant randomized to placebo arm received MK-6096 10 mg) | 83 (1 participant randomized to placebo arm received MK-6096 10 mg)
Completed | 0 | 87 | 82
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-6096 10 mg→No Treatment | MK-6096 10 mg→MK-6096 10 mg | MK-6096 10 mg→Placebo | Total
Number analyzed (Participants) | 12 | 87 | 83 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (6.9) | 55.6 (9.2) | 55.5 (10.3) | 55.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 38 | 36 | 81
  Male | 5 | 49 | 47 | 101

OUTCOME MEASURES:

1. Primary Outcome: Time to Efficacy Failure (TTEF) - Primary Responders
Description: Participants rated their pain twice daily using a 0 to 10 scale with 0=no pain and 10=worst pain you can imagine. The participant's average evening pain intensity scores over the last 3 days of screening period and of run-in period were defined as the run-in baseline score and treatment baseline score, respectively. A primary responder was defined as a participant who had a ≥30% decrease in treatment baseline score relative to run-in baseline score. Efficacy failure was defined as an occurrence of 3 consecutive days, or 4 days in a row with only one day missing and the other 3 days with a daily evening pain intensity score ≥4 and an increase of ≥30% in daily evening pain intensity score relative to treatment baseline score. The time to efficacy failure for primary responders was summarized.
Time Frame: Day 1 of double-blind treatment phase to the first documented efficacy failure (up to 28 days)
Population: All randomized participants (continued into double-blind treatment period) who met criteria as a primary responder.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- MK-6096: Participants who were randomly assigned to receive MK-6096 10 mg during double blind treatment period.
Arm/Group | MK-6096 | Placebo
Number analyzed (Participants) | 37 | 28
Days | NA [NA to NA] — Estimate of median time to efficacy failure is Not Available due to <50% of participants with documented efficacy failure (causing the median to be non-estimable). | NA [NA to NA] — Estimate of median time to efficacy failure is Not Available due to <50% of participants with documented efficacy failure (causing the median to be non-estimable).

2. Secondary Outcome: TTEF - All Responders
Description: Participants rated their pain twice daily using a 0 to 10 scale with 0=no pain and 10=worst pain you can imagine. The participant's average evening pain intensity scores over the last 3 days of screening period and of run-in period were defined as the run-in baseline score and treatment baseline score, respectively. A responder was defined as a participant who had a ≥20% decrease in treatment baseline score relative to run-in baseline score. Efficacy failure was defined as an occurrence of 3 consecutive days, or 4 days in a row with only one day missing and the other 3 days with a daily evening pain intensity score ≥4 and an increase of ≥20% in daily evening pain intensity score relative to treatment baseline score. The time to efficacy failure for responders was summarized.
Time Frame: Day 1 of double-blind treatment phase to the first documented efficacy failure (up to 28 days)
Population: All randomized participants (continued into double-blind treatment period) who met criteria as a responder.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | MK-6096 | Placebo
Number analyzed (Participants) | 47 | 41
Days | NA [NA to NA] — Estimate of median time to efficacy failure is Not Available due to <50% of participants with documented efficacy failure (causing the median to be non-estimable). | NA [NA to NA] — Estimate of median time to efficacy failure is Not Available due to <50% of participants with documented efficacy failure (causing the median to be non-estimable).

3. Secondary Outcome: Change in Pain Intensity Scores - Primary Responders
Description: Participants rated their pain twice daily using a 0 to 10 scale with 0=no pain and 10=worst pain you can imagine. The participant's average evening pain intensity scores over the last 3 days of screening period and of run-in period were defined as the run-in baseline score and treatment baseline score, respectively. A primary responder was defined as a participant who had a ≥30% decrease in treatment baseline score relative to run-in baseline score. The final value was the participant's average evening pain intensity score over the last 3 days of treatment period. The change in the final average evening pain intensity score from treatment baseline was summarized for the primary responders.
Time Frame: End of Single-Blind Period (Baseline) and end of Double-Blind Period
Population: All randomized participants (continued into double-blind treatment period) who met criteria as a primary responder.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-6096 | Placebo
Number analyzed (Participants) | 37 | 28
Score on a Scale | -0.104 [-0.821 to 0.612] | 0.482 [-0.332 to 1.297]
Statistical Analysis 1: Comparison: MK-6096 vs Placebo; Test type: Superiority or Other; p = 0.269, Constrained longitudinal data analysis; terms for treatment, time and treatment-by-time interaction; Difference in Least Squares Means = -0.587, 95% CI 2-sided [-1.637 to 0.464]

4. Secondary Outcome: Change in Pain Intensity Scores - All Responders
Description: Participants rated their pain twice daily using a 0 to 10 scale with 0=no pain and 10=worst pain you can imagine. The participant's average evening pain intensity scores over the last 3 days of screening period and of run-in period were defined as the run-in baseline score and treatment baseline score, respectively. A responder was defined as a participant who had a ≥20% decrease in treatment baseline score relative to run-in baseline score. The final value was the participant's average evening pain intensity score over the last 3 days of treatment period. The change in the final average evening pain intensity score from treatment baseline was summarized for the responders.
Time Frame: End of Single-Blind Period (Baseline) and end of Double-Blind Period
Population: All randomized participants (continued into double-blind treatment period) who met criteria as a responder.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | MK-6096 | Placebo
Number analyzed (Participants) | 47 | 41
Score on a scale | -0.318 [-0.917 to 0.281] | 0.368 [-0.268 to 1.004]
Statistical Analysis 1: Comparison: MK-6096 vs Placebo; Test type: Superiority or Other; p = 0.108, Constrained longitudinal data analysis; terms for treatment, time and treatment-by-time interaction; Difference in Least Squares Means = -0.687, 95% CI 2-sided [-1.527 to 0.154]

5. Primary Outcome: Percentage of Participants Who Experienced 1 or More Adverse Events (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the drug. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an AE.
Time Frame: up to 42 days (up to 14 days for run-in; up to 28 days for active treatment period)
Population: All participants who received at least 1 dose of study drug. One participant who was randomly assigned to placebo for double-blind treatment period actually received MK-6096 10 mg. AEs are reported by treatment received and not by randomly assigned treatment arm.
Measure: Number; unit: Percentage of Participants
Groups:
- MK-6096 10 mg - Run-in Period: Participants who received MK-6096 10 mg during run-in period
- MK-6096 10 Mg-Double Blind Period: Participants who received MK-6096 during double blind treatment period
- Placebo- Double-Blind Period: Participants who received placebo during double-blind treatment period
Arm/Group | MK-6096 10 mg - Run-in Period | MK-6096 10 Mg-Double Blind Period | Placebo- Double-Blind Period
Number analyzed (Participants) | 182 | 88 | 82
Percentage of Participants | 24.7 | 23.9 | 13.4

6. Primary Outcome: Percentage of Participants Who Were Discontinued Form the Study Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the drug. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an AE. Adverse Events that were reported as the cause for discontinuation of the study drug were recorded.
Time Frame: up to 7 days for run-in; up to 14 days for active treatment period)
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-6096 10 mg - Run-in Period | MK-6096 10 Mg-Double Blind Period | Placebo- Double-Blind Period
Number analyzed (Participants) | 182 | 88 | 82
Percentage of Participants | 3.8 | 0.0 | 1.2

ADVERSE EVENTS:
Time Frame: up to 42 days (up to 14 days for run-in; up to 28 days for active treatment period)
Description: All participants who received at least 1 dose of study drug. One participant who was randomly assigned to placebo for double-blind treatment period actually received MK-6096 10 mg. AEs are reported by treatment received and not by randomly assigned treatment arm.
Arm/Group | MK-6096 10 mg - Run-in Period | MK-6096 10 Mg-Double Blind Period | Placebo- Double-Blind Period
Serious Adverse Events (participants affected / at risk) | 3/182 | 0/88 | 1/82
Other Adverse Events (participants affected / at risk) | 0/182 | 0/88 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-6096 10 mg - Run-in Period (N=182) | MK-6096 10 Mg-Double Blind Period (N=88) | Placebo- Double-Blind Period (N=82)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.